CLINICAL TRIAL: NCT06989710
Title: Radicle HealthTM 24: A Randomized, Double-Blind, Placebo-Controlled Direct-to-Consumer Study Assessing the Impact of Health and Wellness Products on Overall Health
Brief Title: Radicle Health 24: A Study of Health and Wellness Products on Overall Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX-P-2405
Record Dates: First submitted 2025-04-14; First posted 2025-05-25 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-06

CONDITIONS: Overall Health

STUDY DESIGN:
Intervention Model Description: Participants will be stratified based on their gender assigned at birth and health outcome score during enrollment, then randomized to one of the study arms. Each participant will have an equal chance of being assigned to any study arm.
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants' assigned study products. Participants are blinded to the study product they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Placebo control 7.1.0 (Placebo Comparator): Health product 7.1.0 - control
  Interventions: Dietary Supplement: Placebo control 7.1.0
- Active product 7.1.1 (Experimental): Health product 7.1.1 - active product 1
  Interventions: Dietary Supplement: Health Active Product 7.1.1 usage
- Active product 7.1.2 (Experimental): Health product 7.1.2 - active product 2
  Interventions: Dietary Supplement: Health Active Product 7.1.2 usage
- Placebo control 7.2.0 (Placebo Comparator): Health product 7.2.0 - control
  Interventions: Dietary Supplement: Placebo control 7.2.0
- Active product 7.2.1 (Experimental): Health product 7.2.1 - active product 1
  Interventions: Dietary Supplement: Health Active Product 7.2.1 usage

INTERVENTIONS:
Dietary Supplement: Placebo control 7.1.0 — Participants will use their placebo control 7.1.0 as directed for a period of 6 weeks.
  Arms: Placebo control 7.1.0
Dietary Supplement: Health Active Product 7.1.1 usage — Participants will use their Radicle Health Active Study Product 7.1.1 as directed for a period of 6 weeks.
  Arms: Active product 7.1.1
Dietary Supplement: Health Active Product 7.1.2 usage — Participants will use their Radicle Health Active Study Product 7.1.2 as directed for a period of 6 weeks.
  Arms: Active product 7.1.2
Dietary Supplement: Placebo control 7.2.0 — Participants will use their placebo control 7.2.0 as directed for a period of 6 weeks.
  Arms: Placebo control 7.2.0
Dietary Supplement: Health Active Product 7.2.1 usage — Participants will use their Radicle Health Active Study Product 7.2.1 as directed for a period of 6 weeks.
  Arms: Active product 7.2.1

SUMMARY:
A randomized, double-blind, placebo-controlled direct-to-consumer study of health and wellness products on overall health

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study conducted with adult participants, residing in the United States.

Eligible participants will (1) endorse a desire for better overall health, (2) have the opportunity for meaningful improvement (at least 30%) in their primary health outcome, and (3) express acceptance in taking a product and not knowing its formulation until the end of the study.

Participants that report a known cardiac dysfunction, liver or kidney disease may be excluded. Participants that report a known contraindication or with well-established, significant safety concerns due to illness will be excluded. Heavy drinkers and those who report they are pregnant, trying to become pregnant, or breastfeeding will be excluded. Participants that report taking medications with a known contraindication or with well-established, significant safety concerns will be excluded.

Self-reported data are collected electronically from eligible participants for 7 weeks. Participant reports of health indicators will be collected at baseline, throughout the active period of study product use, and in a final survey. All study assessments will be electronic; there are no in-person visits or assessments for this real-world evidence study.

ELIGIBILITY:
Inclusion Criteria:

* Adults, at least 21 years of age at the time of electronic consent, inclusive of all ethnicities, races, and gender identities - Assigned sex at birth will determine sex-specific recruitment and surveys (male vs female) employed, when needed
* Resides in the United States
* Endorses better overall health as a primary desire
* Has the opportunity for at least 30% improvement in their primary health outcome
* Expresses a willingness to take a study product and not know the product identity (active or placebo) until the end of the study

Exclusion Criteria:

Report being pregnant, trying to become pregnant, or breastfeeding

* Unable to provide a valid US shipping address and mobile phone number
* Reports current enrollment in another clinical trial
* Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day)
* Unable to read and understand English
* Reports a current and/or recent (up to 3 months ago) major illness and/or surgery that poses a known, significant safety risk.
* Reports a diagnosis of cardiac dysfunction, liver or kidney disease that presents a known contraindication and/or a significant safety risk with any of the study product ingredients.

  o NYHA Class III or IV congestive heart failure, atrial fibrillation, uncontrolled arrhythmias, cirrhosis, end-stage liver disease, stage 3b or 4 chronic kidney disease, or kidney failure
* Reports taking medications that have a well-established moderate or severe interaction, posing a substantial safety risk with any of the study product ingredients.

  o Anticoagulants, antihypertensives, anxiolytics, antidepressants, chemotherapy, immunotherapy, sedative hypnotics, seizure medications, medications that warn against grapefruit consumption, corticosteroids at doses greater than 5 mg per day, diabetic medications, oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection, antipsychotics, MAOIs, or thyroid products
* Reports current use of the primary ingredient(s) and/or similar product(s) to the active study product(s) that may limit the effects of the study products
* Lack of reliable daily access to the internet

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1700 (Actual)
Dates: Start 2025-05-02 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Change in overall health Profile | 7 weeks
  Difference between rates of change over time in overall health score as assessed by Patient Reported Outcome Measurement System (PROMIS) 29+2 Profile (PROPr consists of 7 health domains: physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, cognitive function abilities; PROPr t-score score range = -.022 to 1; higher scores indicate greater overall health)

SECONDARY OUTCOMES:
Minimal clinical importance difference (MCID) in overall health-related quality of life | 7 weeks
  Likelihood of achieving a MCID in digestion-related quality of life, as measured by (PROMIS) 29+2 Profile (PROPr consists of 7 health domains: physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, cognitive function abilities; PROPr t-score score range = -.022 to 1; higher scores indicate greater overall health)
Change in sexual health - female | 7 weeks
  Difference between rates of change over time in sexual health score as assessed by Patient Reported Outcome Measurement System (PROMIS) Brief Profile Sexual Function and Satisfaction Survey [female version consists of 8 health domains: interest in sexual activity (score range = 2-10; higher scores indicate greater interest), vaginal lubrication (score range = 2-10; higher scores indicate better lubrication), vaginal discomfort (score range = 2-10; higher scores indicate more discomfort), vaginal discomfort - labial (score range = 1-5; higher scores indicate more discomfort), vaginal discomfort - clitoral (score range = 1-4; higher scores indicate more discomfort), orgasm ability (score range = 1-5; higher scores indicate more ability), orgasm pleasure (score range = 1-5; higher scores indicate more pleasure), satisfaction with sex life (score range = 2-10; higher scores indicate more satisfaction)]
Change in sexual health - male | 7 weeks
  Difference between rates of change over time in sexual health score as assessed by Patient Reported Outcome Measurement System (PROMIS) Brief Profile Sexual Function and Satisfaction Survey [male version consists of 5 health domains: interest in sexual activity (score range = 2-10; higher scores indicate greater interest), erectile function (score range = 2-10; higher scores indicate better erectile function), orgasm ability (score range = 1-5; higher scores indicate more ability), orgasm pleasure (score range = 1-5; higher scores indicate more pleasure), satisfaction with sex life (score range = 2-10; higher scores indicate more satisfaction)]
Change in GI-related Quality of Life (QOL) | 7 weeks
  Difference between rates of change over time in GI-related QOL as assessed by Digestion-associated QOL Questionnaire (DGLQ) (score range = 0-9; with higher scores corresponding to worse GI-related QOL)
Change in mood (emotion distress-depression) | 7 weeks
  Difference between rates of change over time in emotional distress score as assessed by PROMIS Emotional Distress- Depression 4A (scale 4-20; with higher scores corresponding to greater levels of emotional distress)
Minimal clinically important difference (MCID) in GI-related QOL | 7 weeks
  Likelihood of experiencing minimal clinically important difference in GI-related QOL score as assessed by Digestion-associated QOL Questionnaire (DGLQ) (score range = 0-9; with higher scores corresponding to worse GI-related QOL)
Minimal clinically important difference (MCID) in mood (emotional distress-depression) | 7 weeks
  Likelihood of experiencing minimal clinically important difference in mood score as assessed by PROMIS Emotional Distress- Depression 4A (scale 4-20; with higher scores corresponding to greater levels of emotional distress)
Minimal clinically important difference (MCID) in sexual health - female | 7 weeks
  Likelihood of experiencing minimal clinically important difference in mood score as assessed by PROMIS Brief Profile Sexual Function and Satisfaction Survey [female version consists of 8 health domains: interest in sexual activity (score range = 2-10; higher scores indicate greater interest), vaginal lubrication (score range = 2-10; higher scores indicate better lubrication), vaginal discomfort (score range = 2-10; higher scores indicate more discomfort), vaginal discomfort - labial (score range = 1-5; higher scores indicate more discomfort), vaginal discomfort - clitoral (score range = 1-4; higher scores indicate more discomfort), orgasm ability (score range = 1-5; higher scores indicate more ability), orgasm pleasure (score range = 1-5; higher scores indicate more pleasure), satisfaction with sex life (score range = 2-10; higher scores indicate more satisfaction)]
Minimal clinically important difference (MCID) in sexual health - male | 7 weeks
  Likelihood of experiencing minimal clinically important difference in mood score as assessed by PROMIS Brief Profile Sexual Function and Satisfaction Survey [male version consists of 5 health domains: interest in sexual activity (score range = 2-10; higher scores indicate greater interest), erectile function (score range = 2-10; higher scores indicate better erectile function), orgasm ability (score range = 1-5; higher scores indicate more ability), orgasm pleasure (score range = 1-5; higher scores indicate more pleasure), satisfaction with sex life (score range = 2-10; higher scores indicate more satisfaction)]

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hewlings, Principal Investigator — Radicle Science Inc.
Locations (1):
- Radicle Science, Inc, Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Radicle Science, Inc — http://radiclescience.com